CLINICAL TRIAL: NCT05076695
Title: Neoadjuvant With Trastuzumab, Pyrotinib Plus Palbociclib and Fulvestrant in HER2-positive, ER-positive Breast Cancer
Acronym: NeoTPPF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N032
Record Dates: First submitted 2021-09-18; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Estrogen Receptor-positive Breast Cancer; HER2-positive Breast Cancer
MeSH Terms: interventions — palbociclib; Trastuzumab; pyrotinib; Fulvestrant

STUDY DESIGN:
Intervention Model Description: Patients will enter the single-arm treatment group and they will receive a combination regimen (trastuzumab, pyrotinib, palbociclib plus Fulvestrant, TPPF) as neoadjuvant therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TPPF group (Experimental): Patients will be treated with Trastuzumab, Pyrotinib, Palbociclib plus Fulvestrant(TPPF).
  Interventions: Drug: Palbociclib; Drug: trastuzumab; Drug: pyrotinib; Drug: fulvestrant

INTERVENTIONS:
Drug: Palbociclib — Palbociclib will be given at the dose of 125 mg po q.d. x 21 every 4 weeks (i.e. 1 week rest period for a total of 5 cycles)
Drug: trastuzumab — 8 mg/kg loading dose IV, then 6 mg/kg IV, every 3 weeks for a total of 6 administrations.
Drug: pyrotinib — Pyrotinib 400mg, PO daily, continuously
Drug: fulvestrant — Fulvestrant will be administered according to local prescription guidelines and will be given intramuscle at the dose of 500 mg every 4 weeks (repeat for 5 times) with an additional 500 mg dose given two weeks after the initial dose.

SUMMARY:
This is a prospective Single-arm Study to Investigate the Efficacy and Safety of Neoadjuvant treatment with trastuzumab and pyrotinib plus palbociclib and fulvestrant in HER2-positive, ER-positive breast cancer.

DETAILED DESCRIPTION:
ER+HER2+ breast cancer have low response to single endocrine therapy, however the efficacy was improved when treated with endocrine therapy combined with anti-HER2 target therapy. Palbociclib, to be a CDK4/6 inhibitor, has synergistic with tamoxifen and trastuzumab in ER+/HER2+ cells. In China, there is nearly 40000 new patients with ER+/HER2+ breast cancer every year. The encouraging results in NA-PHER2 study suggested the triple targeting of ER, HER2, and RB1 could be an effective chemotherapy-free treatment strategy in neoadjuvant therapy. However, pertuzumab is very expensive. The investigators plan to replace pertuzumab with pyrotinib. Pyrotinib, a new irreversible pan-Her inhibitor in China pharmaceutical company. The objective is to evaluate the efficacy and safety of Neoadjuvant treatment with trastuzumab and pyrotinib plus palbociclib and fulvestrant (TPPF) in this target population. 37 patients will enter the single-arm treatment group. The participants will receive an association of drugs (trastuzumab, pyrotinib, palbociclib plus Fulvestrant, TPPF) as neoadjuvant therapy. Surgery will be performed not earlier than 14 days and not later than 28 days after the last dose of any of the drugs in the combination. The primary endpoint is the rate of pathological complete response (pCR) defined as ypT0-ypTis ypN0 at surgery. The secondary endpoint include the change in Ki67 expression from baseline and at C2D15 of treatment and at surgery, objective response rate and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 or older than 18;
2. Postmenopausal; Pre-menopausal and peri-menopausal female patients must receive ovarian function inhibitors or ovariectomy concurrently.
3. Have not received chemotherapy or endocrine therapy in the past;
4. Have been confirmed as breast invasive ductal carcinoma by the imaging examination and pathological biopsy;
5. Patients with locally advanced breast cancer, stage IIa-IIIa
6. HER2 status to be centrally confirmed (HER2 3+ of neu amplified)
7. Positive estrogen receptor (ER) > 10%
8. Estimated survival > 12 months;
9. ECOG physical status score before treatment is 0-1 points;
10. The patient has a measurable lesion (according to the standard RECIST 1.1);
11. Willing to cooperate with pre-treatment needle biopsy and neoadjuvant therapy;
12. No serious metastasis, no brain metastasis, no liver metastasis;
13. Normal bone marrow function, blood neutrophils ≥ 1.5x109 / L, hemoglobin ≥ 100g / L, platelets ≥ 100x109 / L;
14. normal liver and kidney function, blood AST≤60U/L, total bilirubin ≤2.5 times of the normal upper limit, and serum creatinine ≤110µmol/L, urea nitrogen ≤7.1mmol/L;
15. No abnormal blood coagulation;
16. Normal heart function, normal ECG and LVEF ≥ 55%;
17. Women of childbearing age are willing to take reliable contraceptive measures during clinical trials, and the serum or urine pregnancy test is negative within 7 days before administration; no coagulation abnormality;
18. Sign the informed consent form (ICF) and voluntarily receive follow-up visits, treatment, laboratory tests and other study procedures as planned.

    -

Exclusion Criteria:

1. Have performed any local or systemic treatment (including chemotherapy, radiotherapy, targeted drug therapy, experimental treatment, etc.) for the breast cancer;
2. Inflammatory breast cancer, bilateral breast cancer or breast cancer with distant metastasis found;
3. Subjects with uncontrolled lung disease, severe infection, active gastrointestinal ulcer, coagulopathy, severe uncontrolled diabetes, connective tissue disease or inhibition of bone marrow function who cannot tolerate neoadjuvant therapy and related therapy;
4. Peripheral neuropathy caused by any factor > 1 degree;
5. Subjects who previously have a history of congestive heart failure, uncontrolled or symptomatic angina, arrhythmia or myocardial infarction, and uncontrollable hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 100 mmHg);
6. Previous extensive radiotherapy
7. Current use or anticipated need for food or drugs that are known strong CYP3A4 (cytochrome P450 3A4) inhibitors or inducers.

   1. Strong CYP3A inhibitors, including, boceprevir, clarithromycin, conivaptan, delavirdine, indinavir, itraconazole, ketoconazole, lopinavir, mibefradil, miconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, suboxone, telaprevir, telithromycin, voriconazole, and grapefruit, grapefruit juice or any product containing grapefruit.
   2. Strong CYP3A inducers, including carbamazepine, phenytoin, primidone, rifampin, rifapentin, and St. John's wort.
8. Breast cancer during the lactation period and gestation period;
9. Reluctance to receive pre-treatment biopsy and neoadjuvant therapy;
10. Psychiatric patients or other factors that cause non-compliance with the treatment;
11. Subjects who are known to have a history of severe allergies to any drug in the treatment regimen; patients who have undergone major surgery or severe trauma within 2 months prior to the first administration; subjects who currently or recently (within 30 days prior to enrolment) have used another investigational drug or participated in another study;
12. Subjects who are known to have infected with human immunodeficiency virus (HIV);
13. Subjects who have other conditions unsuitable for inclusion as considered by investigators, combined with CYP3A4 inhibitors or inducers;
14. Subjects with long QT syndrome or QTc > 470 ms.
15. According to the judgement of the researchers, there are concomitant diseases that seriously endanger the safety of patients or affect the completion of research (including, but not limited to, severe hypertension, severe diabetes, active infections, etc.).
16. Moderate infection occurs within 4 weeks before the first administration (e.g. intravenous drip of antibiotics, antifungal or antiviral drugs according to clinical criteria), fever of unknown origin occurs during the screening period/before the first administration.

    -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2021-10-15 (Estimated); Primary Completion 2023-10-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) | Immediately after the surgery,through study completion, an average of 1 year
  Defined as the absence of any invasive cancer cells in the resected breast specimen and all resected lymph nodes following the completion of neoadjuvant therapy. If there is only carcinoma in situ remains, it can be regarded as pCR.

SECONDARY OUTCOMES:
changes of Ki67 | through study completion, an average of 1 year
  changes of Ki67 from baseline and at cycle2/day 15 and at surgery (approximately 22 weeks after start of neoadjuvant therapy.
objective response rate (ORR) | at the end of the combination treatment, up to 1 year
  The proportion of participants whose best outcome is complete remission or partial remission (according to RECIST1.1)

CONTACTS AND LOCATIONS:
Overall Officials: zhimin U Shao, professor, Principal Investigator — Fudan University Shanghai Cancer Center Shanghai, China, 200032
Locations (1):
- Fudan University Shanghai Cancer Hospital, Shanghai, Shanghai Municipality, China